CLINICAL TRIAL: NCT02113969
Title: Conservative Management of Symptomatic Pelvic Organ Prolapse Using Vaginal Pessaries: Generation of a Standardized Management Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Servicio de Salud Metropolitano Sur Oriente (Other Government)
Collaborators: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SA12I2153
Record Dates: First submitted 2014-04-09; First posted 2014-04-15 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Pelvic Organ Prolapse; Quality of Life
Keywords: Pelvic Organ Prolapse; Quality of Life; Symptoms; Pessary; Treatment
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Pessaries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaginal Pessary (Experimental): Pessary users for at least 12 months
  Interventions: Device: Vaginal Pessary

INTERVENTIONS:
Device: Vaginal Pessary — Pessary fitting session at recruitment, follow up at 1 week, then monthly to complete 1 year follow up. QoL, symptoms and sexual function Surveys will be conducted at recruitment, 6 and 12 month. The absence of bacterial vaginosis (through study of vaginal discharge and pH) will be checked prior to positioning pessary and then each control. At the end of follow up period the success related variables will be determine with a statistical model. This information will be analyzed by an expert panel aiming to identify relevant clinical variables not included. This panel will generate a Standardized Management Protocol for symptomatic pelvic organ prolapse using vaginal pessaries.

SUMMARY:
Genital prolapse is a common condition (up 20%), affecting the quality of life. Treatment can be surgical or conservative using vaginal pessaries. These devices are introduced into the vagina aiming to reduces the prolapse.

Pessaries have shown effectiveness in improving symptoms and quality of life. There are no randomized studies comparing them with surgery. This study design would be difficult to perform, because the inclusion criteria for both treatments are different. There are no currently standard protocols for the use of pessaries. This makes harder to widespread the usage of this conservative treatment.

The aim of the investigators is to identify variables that influence the success of conservative management of genital prolapse at 1 year of follow up. Using these variables and an expert panel opinion the investigators will develop a standardized protocol for pessary management.

Chile has a primary gynecological care system based midwives. Therefore having algorithms for pessaries usage becomes relevant. This algorithm can be implemented with basic training. This would increase the respond capacity, by the health care system to this disease, considering the scarce access to surgery.

The investigators hypothesis is: It is possible to generate a standardized protocol of conservative management of symptomatic genital prolapse in patient's beneficiary of public health system in Santiago, Chile, using pessaries through a prospective cohort study based in the success of these devices with 1 year of follow up, measured with questionnaires of symptoms, quality of life and sexuality

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Pelvic Organ Prolapse
* Commitment to attend controls
* Current negative cervical cytology
* Informed consent signed

Exclusion Criteria:

* Urinary incontinence as the only Pessary Indication
* Vaginal bleeding of undetermined cause
* Unable to return to controls

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Quality of Life changes in pessary users for symptomatic Pelvic Organs Prolapse | 6 months and 12 months
  At baseline, 6 and 12 month the Chilean Version of the P-QoL survey will be applied to describe the QoL changes
Pelvic Floor Disorders symptoms changes in pessary users for symptomatic Pelvic Organs Prolapse | 6 months and 12 months
  At baseline, 6 and 12 month the Chilean Version of the Pelvic Distress Inventory - 20 (PDFI-20) survey will be applied to describe the symptoms changes
Sexual response changes in pessary sexually active women users for symptomatic Pelvic Organs Prolapse | 6 months and 12 months
  At baseline, 6 and 12 month the Chilean Version of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) survey will be applied to describe the Sexually response changes
Subjective impression of improvement after pessary use for symptomatic Pelvic Organs Prolapse | 6 months and 12 months
  At baseline, 6 and 12 month the Patient Global Impression of Improvement (PGI-I) survey will be applied to describe the subjective improvement
Successful usage of pessary | 12 months
  If an enrolled patients is still using the pessary as the treatment for the pelvic organ prolapse will be considered as "successful".
  Risk factors for unsuccessful pessary used will be measure using baseline characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pizarro, MD, Principal Investigator — Complejo Asistencial Dr. Sotero del Rio; Bernardita Blumel, MD, Study Director — Complejo Asistencial Dr. Sotero del Rio; Silvana Gonzalez, Midwife, Study Chair — Complejo Asistencial Dr. Sotero del Rio; Alejandro Pattillo, MD, Study Director — H. Dr. Sotero del Rio; Pontificia Universidad Católica de Chile
Locations (1):
- Unidad de Uroginecologia, Complejo Asistencial Dr. Sotero del Rio, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Derived] Arellano M, Santis-Moya F, Maluenda A, Pattillo A, Blumel B, Pohlhammer D, Gonzalez S, Pizarro-Berdichevsky J. Prevalence of colorectal symptoms and anal incontinence in patients with pelvic organ prolapse attended at an outpatient urogynecology service. Rev Bras Ginecol Obstet. 2024 Mar 15;46:e-rbgo10. doi: 10.61622/rbgo/2024AO10. eCollection 2024. PMID 38765524